CLINICAL TRIAL: NCT00492557
Title: A Phase 3, Randomized, Double-blind Trial to Evaluate Safety, Tolerability, and Immunogenicity of a 13-Valent Pneumococcal Conjugate Vaccine When Administered Concomitantly With Trivalent Inactivated Influenza Vaccine in Healthy Adults 65 Years of Age or Older, Who Are Naive to 23-Valent Pneumococcal Polysaccharide Vaccine
Brief Title: Study Evaluating Safety and Immunogenicity of 13-Valent Pneumococcal Conjugate Vaccine With Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6115A1-3008
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-01

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal Disease; Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13vPnC+TIV Followed by Placebo 1 month later (Experimental)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- Placebo+TIV Followed by 13vPnC 1 month later (Active Comparator)
  Interventions: Biological: 13vPnC + TIV

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — Single 0.5 milliliter (mL) 13-valent pneumococcal conjugate vaccine (13vPnC) and a single 0.5 mL trivalent inactivated influenza vaccine (TIV), administered intramuscularly (IM), followed by a single 0.5 mL vaccine 13vPnC placebo, 1 month later.
  Arms: 13vPnC+TIV Followed by Placebo 1 month later
Biological: 13vPnC + TIV — Single 0.5 mL 13vPnC placebo vaccine and a single 0.5 mL TIV, administered IM, followed by a single 0.5 mL 13vPnC vaccine, 1 month later.
  Arms: Placebo+TIV Followed by 13vPnC 1 month later

SUMMARY:
The 13-valent pneumococcal conjugate vaccine (13vPnC) is being developed for adults to prevent pneumococcal diseases such as meningitis (inflammation of the brain lining), septicemia (blood poisoning), and pneumonia (inflammation of the lungs). As trivalent influenza vaccine (TIV) is frequently given to adults, it is important to show that both vaccines can safely be given together without affecting the immune response (body's ability to protect against disease).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy male or female adults 65 years of age or older.
* Available for the duration of the trial - approximately 2 months.
* No previous vaccination with any pneumococcal vaccine.
* No history of severe adverse reaction associated with a vaccine.
* No allergy to egg proteins (eggs or egg products) and chicken proteins.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1185 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1185 participants were enrolled, of which 1160 were randomized.
Groups:
- 13vPnC+TIV Followed by Placebo 1 Month Later: Single 0.5 milliliter (mL) 13-valent pneumococcal conjugate vaccine (13vPnC) and a single 0.5 mL trivalent inactivated influenza vaccine (TIV), administered intramuscularly (IM), followed by a single 0.5 mL 13vPnC placebo vaccine, 1 month later.
- Placebo+TIV Followed by 13vPnC 1 Month Later: Single 0.5 mL 13vPnC placebo vaccine and a single 0.5 mL TIV, administered IM, followed by a single 0.5 mL 13vPnC, 1 month later.
Period: Overall Study
Arm/Group | 13vPnC+TIV Followed by Placebo 1 Month Later | Placebo+TIV Followed by 13vPnC 1 Month Later
Started | 580 | 580
Vaccinated Dose 1 | 577 | 575
Vaccinated Dose 2 | 560 | 558
Completed | 556 | 557
Not Completed | 24 | 23
Not completed — Subject request | 12 | 11
Not completed — Protocol Violation | 7 | 8
Not completed — Other | 2 | 2
Not completed — Death | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Failed to return | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC+TIV Followed by Placebo 1 Month Later | Placebo+TIV Followed by 13vPnC 1 Month Later | Total
Number analyzed (Participants) | 576 | 575 | 1151
Age Continuous [Mean (Standard Deviation); unit: years] — Data for participants in the safety population (ie. those who received at least 1 dose of study vaccine) are presented. The number of participants equals the number receiving Dose 1 in the Participant Flow section (1152), minus 1 participant in the "13vPnC+TIV followed by placebo 1 month later" group who received a regimen that was not part of the study.
  years | 72.1 (5.6) | 72.1 (5.5) | 72.1 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Data for participants in the safety population (ie. those who received at least 1 dose of study vaccine) are presented. The number of participants equals the number receiving Dose 1 in the Participant Flow section (1152), minus 1 participant in the "13vPnC+TIV followed by placebo 1 month later" group who received a regimen that was not part of the study.
  Participants
    Female | 289 | 290 | 579
    Male | 287 | 285 | 572

OUTCOME MEASURES:

1. Primary Outcome: TIV Comparisons: Percentage of Participants Achieving at Least a 4-fold Increase in the Titer of the Standard Hemagglutination Inhibition Assay (HAI)
Description: Percentage of participants achieving at least a 4-fold increase in the titer of the standard HAI for each influenza virus subtype (A/H1N1, A/H3N2, and B) were compared.
Time Frame: Baseline and 1 month after TIV vaccination
Population: Evaluable immunogenicity population: had participants who adhered to protocol requirements, had valid and determinate assay results, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 13vPnC+TIV: Single 0.5 milliliter (mL) 13-valent pneumococcal conjugate vaccine (13vPnC) and a single 0.5 mL trivalent inactivated influenza vaccine (TIV), administered intramuscularly (IM).
- Placebo+TIV: Single 0.5 mL 13vPnC placebo vaccine and a single 0.5 mL TIV, administered IM.
Arm/Group | 13vPnC+TIV | Placebo+TIV
Number analyzed (Participants) | 549 | 547
Percentage of participants
  Influenza virus subtype: A/H1N1 | 80.3 [76.7 to 83.5] | 78.6 [74.9 to 81.9]
  Influenza virus subtype: A/H3N2 | 58.0 [53.7 to 62.2] | 62.6 [58.4 to 66.6]
  Influenza virus subtype: B | 52.2 [47.9 to 56.4] | 54.0 [49.7 to 58.3]
Statistical Analysis 1: Comparison: 13vPnC+TIV vs Placebo+TIV; Influenza virus subtype: A/H1N1. Primary null hypothesis for each of the influenza virus subtypes is: proportion of participants achieving a 4-fold increase in titer when 13vPnC+TIV were administered concomitantly, minus the proportion of participants achieving a 4-fold increase in titer when TIV was administered alone (with placebo) <= -0.10; Test type: Non-Inferiority or Equivalence — Non-inferiority for a given virus subtype was demonstrated if the lower bound of the 2-sided, 95% confidence interval (CI), computed using the Chan and Zhang procedure, for the difference in proportions (13vPnC+TIV - TIV alone) was greater than -0.10; Percent Difference = 1.7, 95% CI 2-sided [-3.1 to 6.5]
Statistical Analysis 2: Comparison: 13vPnC+TIV vs Placebo+TIV; Influenza virus subtype: A/H3N2. Primary null hypothesis for each of the influenza virus subtypes is: proportion of participants achieving a 4-fold increase in titer when 13vPnC+TIV were administered concomitantly, minus the proportion of participants achieving a 4-fold increase in titer when TIV was administered alone (with placebo) <= -0.10; Test type: Non-Inferiority or Equivalence — Non-inferiority for a given virus subtype was demonstrated if the lower bound of the 2-sided, 95% CI, computed using the Chan and Zhang procedure, for the difference in proportions (13vPnC+TIV - TIV alone) was greater than -0.10; Percent Difference = -4.6, 95% CI 2-sided [-10.4 to 1.3]
Statistical Analysis 3: Comparison: 13vPnC+TIV vs Placebo+TIV; Influenza virus subtype: B. Primary null hypothesis for each of the influenza virus subtypes is: proportion of participants achieving a 4-fold increase in titer when 13vPnC+TIV were administered concomitantly, minus the proportion of participants achieving a 4-fold increase in titer when TIV was administered alone (with placebo) <= -0.10; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Percent Difference = -1.8, 95% CI 2-sided [-7.8 to 4.1]

2. Primary Outcome: 13vPnC Comparisons: Serotype-specific Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentration (GMC)
Description: IgG GMC as measured by enzyme-linked immunosorbent assay (ELISA) and expressed in micrograms per mL (mcg/mL) for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: 1 month after 13vPnC vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Groups:
- 13vPnC: Single 0.5 mL 13vPnC (administered 1 month after single 0.5 mL 13vPnC placebo vaccine and a single 0.5 mL TIV, IM).
Arm/Group | 13vPnC+TIV | 13vPnC
Number analyzed (Participants) | 549 | 547
mcg/mL
  Serotype 1 | 2.52 [2.07 to 3.06] | 3.20 [2.61 to 3.91]
  Serotype 3 | 1.08 [0.94 to 1.24] | 1.15 [1.01 to 1.30]
  Serotype 4 | 2.15 [1.79 to 2.60] | 3.24 [2.65 to 3.96]
  Serotype 5 | 4.74 [4.08 to 5.50] | 6.90 [5.87 to 8.11]
  Serotype 6A | 4.61 [4.00 to 5.31] | 6.10 [5.13 to 7.24]
  Serotype 6B | 6.24 [5.27 to 7.39] | 6.43 [5.33 to 7.76]
  Serotype 7F | 7.63 [6.50 to 8.96] | 9.04 [7.58 to 10.79]
  Serotype 9V | 4.97 [4.19 to 5.91] | 6.21 [5.27 to 7.33]
  Serotype 14 | 8.95 [7.33 to 10.95] | 12.44 [9.94 to 15.57]
  Serotype 18C | 8.88 [7.55 to 10.45] | 11.07 [9.40 to 13.04]
  Serotype 19A | 11.93 [10.23 to 13.92] | 17.10 [14.54 to 20.10]
  Serotype 19F | 4.78 [4.00 to 5.71] | 7.39 [6.02 to 9.08]
  Serotype 23F | 5.82 [4.74 to 7.14] | 6.11 [4.97 to 7.50]
Statistical Analysis 1: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 1. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — The criterion upon which to declare non-inferiority was the lower bound of the 2-sided, 95% CI for the geometric mean ratio greater than 0.5 (2-fold criterion); Ratio of GMCs = 0.79, 95% CI 2-sided [0.60 to 1.04] — CIs for the ratio were back transformations of the CIs based on the Student t distribution for the mean difference of the logarithmically transformed assay results
Statistical Analysis 2: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 3. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.94, 95% CI 2-sided [0.78 to 1.13] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 4. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.66, 95% CI 2-sided [0.51 to 0.87] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 5. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.69, 95% CI 2-sided [0.55 to 0.86] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 6A. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.76, 95% CI 2-sided [0.61 to 0.94] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 6B. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.97, 95% CI 2-sided [0.75 to 1.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 7F. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.84, 95% CI 2-sided [0.67 to 1.07] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 9V. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.80, 95% CI 2-sided [0.63 to 1.02] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 14. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.72, 95% CI 2-sided [0.53 to 0.97] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 18C. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.80, 95% CI 2-sided [0.64 to 1.01] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 19A. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.70, 95% CI 2-sided [0.56 to 0.87] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 19F. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.65, 95% CI 2-sided [0.49 to 0.85] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 23F. The primary null hypothesis was: the log of the GMC in the group receiving 13vPnC and TIV concomitantly, minus the log of the GMC in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of GMCs = 0.95, 95% CI 2-sided [0.71 to 1.27] — [estimate comment as in outcome 2, analysis 1]

3. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions
Description: Local reactions were reported using an electronic diary. Pain was scaled as Any; Mild (awareness but easily tolerated); Moderate (discomfort enough to interfere with usual activity) and Severe (incapacitating the usual activity). Redness and swelling were scaled as Any; Mild (2.5 cm to 5.0 cm); Moderate (5.1 to 10.0 cm)and Severe (> 10.0 cm). Limitation in arm movement were scaled as Any; Mild (some limitation); Moderate (unable to move above head but able to move above shoulder) and Severe (unable to move above shoulder).
Time Frame: Days 1 through 14 after 13vPnC vaccination
Population: Safety population: included all participants who received at least 1 dose of study vaccine. n=number of participants at each timepoint, in each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+TIV | 13vPnC
Number analyzed (Participants) | 577 | 558
percentage of participants
  Redness: Any (n= 440, 432) | 16.6 [-0.4 to 9.0] | 12.3 [-0.4 to 9.0]
  Redness: Mild (n= 438, 432) | 14.4 [0.3 to 9.1] | 9.7 [0.3 to 9.1]
  Redness: Moderate (n= 433, 424) | 6.0 [-3.4 to 3.1] | 6.1 [-3.4 to 3.1]
  Redness: Severe (n= 429, 420) | 0.7 [-1.8 to 1.2] | 1.0 [-1.8 to 1.2]
  Swelling: Any (n= 441, 431) | 13.8 [-0.7 to 8.0] | 10.2 [-0.7 to 8.0]
  Swelling: Mild (n= 440, 430) | 11.8 [-0.3 to 7.7] | 8.1 [-0.3 to 7.7]
  Swelling: Moderate (n= 432, 423) | 4.2 [-3.7 to 2.1] | 5.0 [-3.7 to 2.1]
  Swelling: Severe (n= 428, 420) | 0.2 [-0.7 to 1.3] | 0.0 [-0.7 to 1.3]
  Pain: Any (n= 480, 470) | 40.0 [-9.7 to 3.0] | 43.4 [-9.7 to 3.0]
  Pain: Mild (n= 470, 462) | 34.3 [-9.8 to 2.6] | 37.9 [-9.8 to 2.6]
  Pain: Moderate (n= 447, 442) | 14.8 [-9.9 to 0.1] | 19.7 [-9.9 to 0.1]
  Pain: Severe (n= 429, 421) | 1.4 [-3.4 to 0.8] | 2.6 [-3.4 to 0.8]
  Limitation of arm movement: Any (n= 445, 432) | 13.9 [-5.6 to 3.8] | 14.8 [-5.6 to 3.8]
  Limitation of arm movement: Mild (n= 444, 432) | 13.1 [-4.9 to 4.2] | 13.4 [-4.9 to 4.2]
  Limitation of arm movement:Moderate (n= 430, 420) | 1.4 [-1.2 to 2.2] | 1.0 [-1.2 to 2.2]
  Limitation of arm movement: Severe (n= 429, 420) | 1.9 [-1.4 to 2.4] | 1.4 [-1.4 to 2.4]
  Any local reaction (n= 488, 470) | 46.9 [-6.0 to 6.7] | 46.6 [-6.0 to 6.7]

4. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events
Description: Systemic events (Any fever >= 38 degrees Celsius [C]), fatigue, headache, chills, rash, vomiting, decreased appetite, new muscle pain, any aggravated muscle pain, new joint pain or any aggravated joint pain. Participants may be presented in more than one category.
Time Frame: Days 1 through 14 after 13vPnC vaccination
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC+TIV | 13vPnC
Number analyzed (Participants) | 577 | 558
Percentage of participants
  Fever >=38 degreesC but <38.5 degreesC (n=434,423) | 3.0 [-2.5 to 2.3] | 3.1 [-2.5 to 2.3]
  Fever >=38.5 degreesC but <39 degreesC (n=430,421) | 1.4 [-1.2 to 2.2] | 1.0 [-1.2 to 2.2]
  Fever >=39degreesC but <=40.0degreesC (n=428,420) | 0.0 [-0.9 to 0.9] | 0.0 [-0.9 to 0.9]
  Fever >40.0 degrees C (n= 429, 422) | 1.4 [-0.8 to 2.4] | 0.7 [-0.8 to 2.4]
  Fatigue (n= 476, 456) | 37.4 [2.8 to 14.9] | 28.5 [2.8 to 14.9]
  Headache (n= 472, 449) | 32.6 [2.1 to 13.8] | 24.7 [2.1 to 13.8]
  Chills (n= 443, 429) | 13.8 [0.4 to 9.0] | 9.1 [0.4 to 9.0]
  Rash (n= 433, 427) | 6.9 [-3.3 to 3.6] | 6.8 [-3.3 to 3.6]
  Vomiting (n= 432, 424) | 3.0 [-0.7 to 3.6] | 1.7 [-0.7 to 3.6]
  Decreased appetite (n= 450, 434) | 16.9 [1.0 to 10.2] | 11.3 [1.0 to 10.2]
  New muscle pain (n= 468, 448) | 26.9 [-2.2 to 9.1] | 23.4 [-2.2 to 9.1]
  Any aggravated muscle pain (n= 454, 439) | 18.7 [-1.2 to 8.7] | 15.0 [-1.2 to 8.7]
  New joint pain (n= 452, 435) | 16.2 [0.1 to 9.2] | 11.5 [0.1 to 9.2]
  Any aggravated joint pain (n= 452, 428) | 15.7 [2.7 to 11.4] | 8.6 [2.7 to 11.4]
  Any systemic event (n= 510, 488) | 60.2 [5.4 to 17.8] | 48.6 [5.4 to 17.8]

5. Post Hoc Outcome: 13vPnC Comparisons: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT)
Description: Pneumococcal OPA GMTs for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of a subset of participants using a microcolony OPA (mcOPA) assay.
Time Frame: 1 month after 13vPnC vaccination
Population: Evaluable immunogenicity population: had participants who adhered to protocol requirements, had valid and determinate assay results, and had no major protocol violations. n= number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | 13vPnC+TIV | 13vPnC
Number analyzed (Participants) | 259 | 255
Geometric mean titers
  Serotype 1 (n= 256, 255) | 88 [71.1 to 108.3] | 95 [76.8 to 117.9]
  Serotype 3 (n= 235, 237) | 46 [37.9 to 56.1] | 51 [41.7 to 61.7]
  Serotype 4 (n= 247, 245) | 997 [766.3 to 1296.0] | 1486 [1174.7 to 1879.8]
  Serotype 5 (n= 245, 234) | 124 [97.3 to 158.8] | 112 [85.1 to 146.3]
  Serotype 6A (n= 250, 252) | 1220 [950.6 to 1566.7] | 1597 [1256.4 to 2030.3]
  Serotype 6B (n= 259, 248) | 1564 [1239.4 to 1973.9] | 2017 [1564.8 to 2599.9]
  Serotype 7F (n= 246, 248) | 607 [444.2 to 828.8] | 835 [619.9 to 1123.9]
  Serotype 9V (n= 247, 242) | 477 [348.5 to 652.7] | 723 [528.1 to 988.9]
  Serotype 14 (n= 247, 236) | 975 [781.6 to 1215.5] | 1088 [858.4 to 1379.1]
  Serotype 18C (n= 250, 244) | 1158 [909.5 to 1475.1] | 1415 [1122.0 to 1785.8]
  Serotype 19A (n= 251, 247) | 445 [365.1 to 542.1] | 539 [427.8 to 679.7]
  Serotype 19F (n= 247, 242) | 378 [295.8 to 483.8] | 467 [360.7 to 605.1]
  Serotype 23F (n= 252, 242) | 245 [180.2 to 332.4] | 295 [217.9 to 400.8]
Statistical Analysis 1: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 1. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — The criterion upon which to declare non-inferiority was if the lower limit of the 2-sided 95%CI for the GMT ratios, (13vPnC+TIV relative to 13vPnC administered 1 month after TIV+placebo) was greater than 0.5 (2-fold criterion); GMT Ratio = 0.9, 95% CI 2-sided [0.68 to 1.24] — 2-sided 95% CIs for the GMT ratio were calculated by back transformations of the 95% CIs based on the Student t distribution for the mean difference of the logarithmically transformed assay results
Statistical Analysis 2: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 3. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.9, 95% CI 2-sided [0.69 to 1.20] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 4. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.7, 95% CI 2-sided [0.47 to 0.95] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 5. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 1.1, 95% CI 2-sided [0.77 to 1.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 6A. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.54 to 1.08] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 6B. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.55 to 1.09] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 7F. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.7, 95% CI 2-sided [0.47 to 1.12] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 9V. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.7, 95% CI 2-sided [0.42 to 1.03] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 14. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.9, 95% CI 2-sided [0.65 to 1.24] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 18C. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.59 to 1.14] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 19A. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.61 to 1.12] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 19F. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.57 to 1.16] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC+TIV vs 13vPnC; Serotype 23F. The primary null hypothesis was: the log of the GMT in the group receiving 13vPnC + TIV minus the log of the GMT in the group receiving 13vPnC alone (1 month after TIV) <= -0.693; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.54 to 1.27] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: AEs/SAEs recorded from signing of informed consent form to completion of study (Visit 3).Participants recorded in the e-diary their local reactions,systemic events & use of antipyretic & pain medication (Day 1-Day 14 after study vaccine administration).
Description: SAEs were grouped by organ system, with number and frequency of events summarized. Non-serious AEs were summarized in a similar manner and included solicited AEs collected in the e-diary (systematic assessment) and unsolicited events collected on the case report form at each visit (non-systematic assessment).
Groups:
- 13vPnC+TIV: Single 0.5 mL 13vPnC and a single 0.5 mL TIV, administered IM.
- Placebo: Single 0.5 mL 13vPnC placebo vaccine (administered 1 month after a single 0.5 mL 13vPnC and a single 0.5 mL TIV, IM [13vPnC + TIV]).
- 13vPnC: Single 0.5 mL 13vPnC (administered 1 month after single 0.5 mL 13vPnC placebo vaccine and a single 0.5 mL TIV, IM [Placebo + TIV]).
Arm/Group | 13vPnC+TIV | Placebo | Placebo+TIV | 13vPnC
Serious Adverse Events (participants affected / at risk) | 4/576 | 8/559 | 0/575 | 5/558
Other Adverse Events (participants affected / at risk) | 307/576 | 194/559 | 256/575 | 237/558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC+TIV (N=576) | Placebo (N=559) | Placebo+TIV (N=575) | 13vPnC (N=558)
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Endoscopy small intestine (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC+TIV (N=576) | Placebo (N=559) | Placebo+TIV (N=575) | 13vPnC (N=558)
Redness (any) (Skin and subcutaneous tissue disorders) | 73/440 | 6/393 | 11/433 | 53/432 — Redness (any) = present at site of vaccination
Redness (mild) (Skin and subcutaneous tissue disorders) | 63/438 | 6/393 | 6/433 | 42/432 — Redness (mild) = 2.5 to 5.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 26/433 | 0/392 | 5/431 | 26/424 — Redness (moderate) = 5.1 to 10.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 3/429 | 0/392 | 0/431 | 4/420 — Redness (severe) = >10.0 cm
Swelling (any) (Skin and subcutaneous tissue disorders) | 61/441 | 4/394 | 12/435 | 44/431 — Swelling (any) = present at site of vaccination
Swelling (mild) (Skin and subcutaneous tissue disorders) | 52/440 | 4/394 | 9/434 | 35/430 — Swelling (mild) = 2.5 to 5.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 18/432 | 1/393 | 5/433 | 21/423 — Swelling (moderate) = 5.1 to 10.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 1/428 | 0/392 | 1/431 | 0/420 — Swelling (severe) = >10.0 cm
Pain (any) (Skin and subcutaneous tissue disorders) | 192/480 | 40/411 | 45/445 | 204/470 — Pain (any) = present at site of vaccination
Pain (mild) (Skin and subcutaneous tissue disorders) | 161/470 | 33/408 | 40/443 | 175/462 — Pain (mild) = awareness of symptoms but easily tolerated
Pain (moderate) (Skin and subcutaneous tissue disorders) | 66/447 | 10/397 | 14/437 | 87/442 — Pain (moderate) = discomfort enough to cause interference with usual activity
Pain (severe) (Skin and subcutaneous tissue disorders) | 6/429 | 0/392 | 0/431 | 11/421 — Pain (severe) = unable to move above shoulder
Limitation of arm movement (any) (Skin and subcutaneous tissue disorders) | 62/445 | 20/397 | 26/440 | 64/432 — Limitation of arm movement (any) = present
Limitation of arm movement (mild) (Skin and subcutaneous tissue disorders) | 58/444 | 17/397 | 26/440 | 58/432 — Limitation of arm movement (mild) = some limitation
Limitation of arm movement (moderate) (Skin and subcutaneous tissue disorders) | 6/430 | 4/393 | 1/432 | 4/420 — Limitation of arm movement (moderate) = unable to move above head but able to move above shoulder
Limitation of arm movement (severe) (Skin and subcutaneous tissue disorders) | 8/429 | 4/392 | 0/431 | 6/420 — Limitation of arm movement (severe) = unable to move above shoulder
Fever ≥ 38 degrees C but < 38.5 degrees C (General disorders) | 13/434 | 8/398 | 8/434 | 13/423
Fever ≥ 38.5 degrees C but < 39 degrees C (General disorders) | 6/430 | 4/394 | 5/433 | 4/421
Fever ≥ 39 degrees C but ≤ 40.0 degrees C (General disorders) | 0/428 | 3/394 | 1/431 | 0/420
Fever > 40.0 degrees C (General disorders) | 6/429 | 4/393 | 10/438 | 3/422
Fatigue (General disorders) | 178/476 | 120/434 | 154/483 | 130/456
Headache (General disorders) | 154/472 | 114/436 | 139/468 | 111/449
Chills (General disorders) | 61/443 | 32/404 | 40/440 | 39/429
Rash (General disorders) | 30/433 | 10/397 | 15/436 | 29/427
Vomiting (General disorders) | 13/432 | 12/398 | 15/437 | 7/424
Decreased appetite (General disorders) | 76/450 | 58/415 | 66/452 | 49/434
New muscle pain (General disorders) | 126/468 | 47/413 | 76/456 | 105/448
Any aggravated muscle pain (General disorders) | 85/454 | 44/410 | 63/449 | 66/439
New joint pain (General disorders) | 73/452 | 45/408 | 59/451 | 50/435
Any aggravated joint pain (General disorders) | 71/452 | 45/407 | 58/447 | 37/428
Arrhythmia (Cardiac disorders) | 1 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 2 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 2 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Sensation of foreign body (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 8 | 9
Nasopharyngitis (Infections and infestations) | 7 | 10 | 6 | 8
Localised infection (Infections and infestations) | 1 | 2 | 2 | 0
Cystitis (Infections and infestations) | 1 | 2 | 1 | 5
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 4
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 3
Enterovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1 | 3
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Total lung capacity decreased (Investigations) | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Nephrocalcinosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Dental prosthesis user (Social circumstances) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 8 | 3 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.